CLINICAL TRIAL: NCT03945383
Title: Clinical Investigation of Safety and Efficacy of the Emerald IPL Device for Hair Reduction for the Extension of Its Intended Use to Face and to Skin Type V Population
Brief Title: Clinical Investigation of Safety and Effectiveness of Emerald IPLdevice
Acronym: Emerald
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PC-BEA-Emerald STV&Face-10560
Record Dates: First submitted 2019-04-29; First posted 2019-05-10 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Hair Removal
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: All enrolled subjects will be treated with the investigational device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment with IPL device (Experimental): The Emerald IPL device is applied by the Investigator or designee to the right and left side of the body. Treatment areas are 2x4 cm2 for the leg and bikini line areas. The entire axilla and face (upper lip) area will be treated due to the small area involved.
  Interventions: Device: Treatment with IPL device

INTERVENTIONS:
Device: Treatment with IPL device — Treatment with IPL device

SUMMARY:
Prospective, multi-center, single-arm, single blinded (Philips hair counter) study in healthy women of skin types I up to and including V.

Safety and efficacy of hair removal with the Emerald IPL-device will be investigated for treatment in face of subjects with ST I - IV and for treatment in face, axilla, bikini area, and legs of subjects with ST V.

In-clinic, the study subjects will undergo twelve IPL-treatments bilaterally at the qualified areas (face and / or axilla, bikini line, and legs) with the Emerald IPL device applied by a device operator.

Hair re-growth in each area will be evaluated separately and across all skin types.

After the 4 bi-weekly treatments, one follow-up visit will be organized two weeks after the 4th treatment. After the completion of the full treatment cycle (12 treatments), subjects will be followed for 1 and 3 months (short-term follow-up) and for 6, 9 and 12 months (long-term follow up).

DETAILED DESCRIPTION:
Hair grows in cyclic phases: anagen, catagen and telogen. These phases impact on how the process of light-based hair removal works. The hair grows during the anagen phase, which has the longest duration in the hair growth cycle. Hair growth ends with the transition from anagen into the catagen phase, a short transition phase to prepare for the resting phase, the telogen, which ends with shedding of the hair and the start of the hair growth cycle. During telogen phase, the hair follicle remains inactive. Each hair follicle is independent and goes through the growth cycle at different times. As presented in table 5 [11], the duration of the growth cycle of the upper lip, axilla and bikini line are different from that of the legs. In general, the telogen and anagen phase's durations of the cycle are longest for the legs (i.e., 24 and 16 weeks, respectively) and the shortest for upper lip (i.e. 6 weeks for both phases). Therefore, hair response to the IPL treatment will be evaluated by body area.

The efficacy of permanent hair reduction will be measured following the definition of permanent hair reduction according to the FDA as follows: "Permanent hair reduction is defined as the long-term, stable reduction in the number of hairs re-growing after a treatment regime, which may include several sessions. The number of hairs re-growing must be stable over time greater than the duration of the complete growth cycle of hair follicles, which varies from four to twelve months according to body location. Permanent hair reduction does not necessarily imply the elimination of all hairs in the treatment area."

In an attempt to promote permanent hair reduction, the aim is to expose all hairs at least once to an IPL flash and therefore treatment will cover the full duration of a hair growth cycle). The longest relevant full hair growth cycle is on the legs (40 weeks, excluding approximately 2 weeks for the catagen phase). Therefore, a treatment duration of 10 months (approximately 38weeks) has been selected: a full IPL treatment cycle consists of 4 initial treatments, once every 2 weeks, followed by 8 maintenance (monthly) treatments, once every 4 weeks. The hair growth cycle on face (upper lip) is the shortest (12 weeks, 6 weeks in anagen, 6 weeks in telogen phases). The initial treatments in 2 weeks interval are expected to be most beneficial for face treatment.

For this study, there are two cohorts for enrollment:

1. Subjects with Skin Type I-IV for treatment of Face only. (N=53)
2. Subjects with Skin Type V for treatment of all body areas: Face, Axilla, Bikini line and leg. (N=19)

The visits are as follows:

Screening Visit: The volunteers are screened to identify subjects who meet all of the inclusion and none of the exclusion criteria. Device settings are selected based on skin tone and comfort evaluation..

Visits 1-4 (TX1-TX4): Four treatments and the collection of safety and efficacy data are scheduled to occur every 2 weeks/ 14 days; Visits 5 (Initial Treatment 2wk Follow-up): Safety and efficacy data are collected 2 weeks/ 14 days after 4th treatment to demonstrate hair removal performance 8 weeks after baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing to provide informed consent
2. Are healthy female subjects, in age of 18-65 years
3. Have natural body hair color that is dark blonde, brown or black in the designated treatment areas

   3.1. Subjects of ST I-IV - Face group:

   3.1.1 Have Fitzpatrick Skin Type I, II, III, or IV

   3.1.2 Measure melanin value ≤ 375 in the qualifying treatment areas bilateral on upper lip (face)

   3.1.3. Have a minimum of 10 hairs in the 1x2cm2 qualifying treatment areas bilateral on upper lip (face), by visual inspection

   3.2. Subjects of ST V - All body area group:

   3.2.1. Have Fitzpatrick Skin Type V

   3.2.2. Measure melanin value ≤ 553 in the qualifying treatment areas bilateral on upper lip (face), axilla, bikini line, and leg

   3.2.3. Have a minimum of 10 hairs in the 1x2cm2 qualifying treatment areas bilateral on upper lip (face), by visual inspection

   3.2.4.Have a minimum of 24 hairs in each of the 2x4cm2 qualifying treatment areas bilateral on axilla, bikini line, and leg, by visual inspection
4. Be either post-menopausal or surgically sterilized, or using a medically acceptable form of birth control (e.g., oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide or abstinence, etc.).
5. Be willing to participate in all study visits
6. Be willing to refrain from deliberate exposure to strong sun, products or procedures that would cause the skin to become darker in the designated treatment areas during the treatment phase
7. Be willing to refrain from the use of hair growth inhibitors/accelerators during the course of the study
8. Be willing to refrain from waxing, depilating or epilating of the axilla, bikini line, leg, and face
9. Be willing to refrain from using aspirin or NSAIDs (e.g. acetaminophen, ibuprofen, etc.) within 5 days prior to and 5 days after treatment(s) -

Exclusion Criteria:

1. Have natural body hair color that is white, light blond, or red in the designated treatment areas

   1.1. Subjects of ST I to IV - Face group:

   1.1.1. Have Fitzpatrick Skin Type V or VI

   1.1.2. Measure melanin value higher than 375 in the qualifying treatment areas bilateral on upper lip

   1.1.3. Have fewer than 2 qualifying treatment areas on bilateral on upper lip (face)

   1.2. Subjects of ST V - All body area group:

   1.2.1. Have Fitzpatrick Skin Type I, II, III, IV, or VI

   1.2.2. Measure melanin value higher than 553 in any of the qualifying treatment areas bilateral on the body

   1.2.3. Have fewer than 8 qualifying treatment areas bilateral: 2 in face, 2 in axilla, 2 on bikini line, and 2 on legs
2. Have a malignant or pre-malignant pigment in the area to be treated
3. Have scarring or infection of the area to be treated
4. Have a known history of photosensitivity or use of medication known to induce photosensitivity
5. Are currently pregnant or lactating or planning be become pregnant in the period of the study, per subject report
6. Are currently on a daily dose of aspirin or NSAIDs (e.g. acetaminophen, ibuprofen, etc.) or have taken aspirin and/or NSAIDs within 5 days prior to treatment that would reduce or increase the sensation of pain
7. Are not willing to abstain from the use of products or light exposure that would induce tanning in the treatment areas during the IPL treatment period (first 10 months)
8. Have a history of immunosuppressive disease (including HIV infection or AIDS)
9. Are on a anticoagulative medication or thromboembolic condition
10. Have taken any form of isotretinoin (such as Accutane or Roaccutane etc.) in the last six months
11. Have an active implantable device such as a pacemaker, neurostimulator or internal defibrillator
12. Have used waxing or other methods of root hair removal, or photo-epilation in the areas to be treated within 6 months prior to treatment
13. Have been exposed to strong sunlight or an artificial tanning machine in the area to be treated within 4 weeks of enrolment
14. Have a tattoo(s), warts, moles, benign skin lesions, dark pigmented areas, permanent make-up etc. in the areas to be treated.
15. Have eczema, psoriasis, lesions, open wounds or any skin affliction in the areas to be treated
16. Have a history of keloid scar formation
17. Have a history of herpes outbreaks in the areas to be treated
18. Have a history of photosensitive epilepsy
19. Have a condition related to hormonal changes like polycystic ovarian syndrome (PCOS) or taking drugs leading to hormonal changes resulting in excessive hair growth like hirsutism or idiopathic hirsutism
20. Have diabetes, or metabolic disease that affects hair growth
21. Taking immunosuppressive medication(s)
22. Have a disease related to photosensitivity, such as polymorphic light eruption (PMLE), solar urticaria, porphyria etc.
23. Have a history of skin cancer, including past basal cell carcinoma and/or squamous cell carcinoma in the areas to be treated
24. Have a history of any radiation therapy in any of the areas to be treated
25. Have history of radiation therapy in non-treatment areas within 5 years
26. Have a history of chemotherapy
27. Have used hair growth inhibitors and/or accelerators within 6 months preceding enrolment
28. Have had laser or electrolysis treatment for the removal of hair in the areas to be treated within the last year
29. Have natural body hair colors of white, grey, light to mid-blond, or red in the areas to be treated
30. Have bleaching of their body hair in the areas to be treated 6 months prior to study enrolment
31. Have shaved the areas to be treated within 7 days prior to study enrolment
32. Participating in other clinical studies prior to, or concurrently with this study, that could be deemed to interfere with full and complete participation in this study - as determined by the site investigator.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with at least 30% hair reduction relative to baseline at 8 and 10 weeks after baseline and at 1 and 3 months after last treatment | approximately 13 months
  Efficacy of the device will be measured by evaluating the proportion of subjects with >= 30% hair reduction on the face, axilae, bikini area and legs following the intensive treatment phase at 8 and 10 weeks as well as during short term follow up of 1 month and 3 months after the last treatment.

SECONDARY OUTCOMES:
Safety will be measured by proportion of treatment-emerged, anticipated adverse events, non-anticipated adverse events, serious adverse events and other related reasons for discontinuation. | Approximately 22 months
  The primary safety endpoints include the treatment-emerged, anticipated adverse events, non-anticipated adverse events, serious adverse events and reasons for discontinuation during the treatment of the face, axilae, bikini area and legs with the device as well as during the follow-up period.
Assessment of the subjective satisfaction with the treatment results of the Emerald IPL device for removal of unwanted hair on face, axillae, bikini area, and legs: 5-point Likert satisfaction scale | Approximately 22 months
  Percent of top-two category answers of 5-point Likert satisfaction scale in assessment of subjective satisfaction with the treatment results in all body areas.
Assessment of the acceptance of the Emerald IPL devices for removal of unwanted hair in each body area: Percent of top-two category answers in assessment of acceptance | Approximately 22 months
  Percent of top-two category answers in assessment of acceptance of hair reduction, skin smoothness, and comfort after treatment with Philips investigational IPL devices in all body areas.
Proportion of subjects with at least 30% hair reduction relative to baseline at 6, 9 and 12 months post-final treatment per body area. | Approximately 22 months
  Efficacy of the device will be measured by evaluating the proportion of subjects with >= 30% hair reduction on the face, axilae, bikini area and legs during the long term follow up of 1 month and 3 months after the last treatment.

OTHER OUTCOMES:
Exploratory Endpoint | Approximately 18 months
  Percent of subjects with the same device setting as Setting Indication by STS device and device setting as result of Test Flash or as result of skin type self-assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Rupal Trivedi, M.D., Principal Investigator — Great Lakes Clinical Trials; David Pariser, M.D., Principal Investigator — Virginia Clinical Research
Locations (3):
- United States (3):
  - My Community Research Center, Miami, Florida
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Virginia Clinical Research, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altshuler GB, Anderson RR, Manstein D, Zenzie HH, Smirnov MZ. Extended theory of selective photothermolysis. Lasers Surg Med. 2001;29(5):416-32. doi: 10.1002/lsm.1136. PMID 11891730
- [Background] Ravnbak MH. Objective determination of Fitzpatrick skin type. Dan Med Bull. 2010 Aug;57(8):B4153. PMID 20682135
- [Background] Shamsuddin K et. al, The reliability of Fitzpatrick Skin Type Chart Comparing to Mexameter (Mx 18) in measuring skin color among first trimester, Malaysian Journal of Public Health Medicine 2016, Vol. 16 (3): 59-65
- [Background] Gold MH, Bell MW, Foster TD, Street S. Long-term epilation using the EpiLight broad band, intense pulsed light hair removal system. Dermatol Surg. 1997 Oct;23(10):909-13. doi: 10.1111/j.1524-4725.1997.tb00746.x. PMID 9357500
- [Background] Gold MH, Bell MW, Foster TD, Street S. One-year follow-up using an intense pulsed light source for long-term hair removal. J Cutan Laser Ther. 1999 Sep;1(3):167-71. doi: 10.1080/14628839950516823. PMID 11360413
- [Background] Dierickx CC. Hair removal by lasers and intense pulsed light sources. Dermatol Clin. 2002 Jan;20(1):135-46. doi: 10.1016/s0733-8635(03)00052-4. PMID 11859588
- [Background] Thaysen-Petersen D, Bjerring P, Dierickx C, Nash JF, Town G, Haedersdal M. A systematic review of light-based home-use devices for hair removal and considerations on human safety. J Eur Acad Dermatol Venereol. 2012 May;26(5):545-53. doi: 10.1111/j.1468-3083.2011.04353.x. Epub 2011 Nov 30. PMID 22126235
- [Background] Town G, Ash C, Dierickx C, Fritz K, Bjerring P, Haedersdal M. Guidelines on the safety of light-based home-use hair removal devices from the European Society for Laser Dermatology. J Eur Acad Dermatol Venereol. 2012 Jul;26(7):799-811. doi: 10.1111/j.1468-3083.2011.04406.x. Epub 2012 Jan 3. PMID 22211702
- [Background] Fitzpatrick TB. The validity and practicality of sun-reactive skin types I through VI. Arch Dermatol. 1988 Jun;124(6):869-71. doi: 10.1001/archderm.124.6.869. No abstract available. PMID 3377516